CLINICAL TRIAL: NCT01355419
Title: Evaluation of Sleep Schedules Modifications in Moderate to Severe Sleep Apnea Patients Treated by nCPAP
Brief Title: Sleep Schedules Modifications in Sleep Apnea Patients Treated by nCPAP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, chef de clinique adjoint, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: AK/10-07-45/3912
Record Dates: First submitted 2011-05-06; First posted 2011-05-18 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP; actigraphy; sleep; physical activity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obstructive sleep apnea, CPAP: moderate to severe obstructive sleep apnea requiring CPAP therapy

SUMMARY:
In Obstructive sleep apnea (OSA) patients, sleep is disrupted and sleep quality is very poor. The investigators can suppose that with continuous positive airway pressure (CPAP) therapy, there is an improvement in sleep quality, such that patients need less sleep to be fit. Sleep schedules on mid term periods in OSA patients under CPAP therapy has not been studied. The investigators have planned to study sleep schemes before and after CPAP therapy in moderate to severe sleepy OSA patients.

DETAILED DESCRIPTION:
In Obstructive sleep apnea (OSA) patients, sleep is disrupted and sleep quality is very poor. The investigators can suppose that with CPAP therapy, there is an improvement in sleep quality, such that patients need less sleep to be fit. Patients often report this fact, but it has not been objectivated.

Sleep schedules on mid term periods in OSA patients under CPAP therapy has not been studied. The investigators have planned to study sleep schemes before and after CPAP therapy in moderate to severe sleepy OSA patients. Sleep schemes and physical activity will be studied with actigraphy.

Study Design : prospective study. Number of patients supposed to be studied: 190

Methods:

Patients Ø OSA patients assessed by polysomnography, showing apnea-hypopnea index > 20, and Epworth Sleepiness Scale Score(ESS) >10 Ø Indication of CPAP therapy

Initial Evaluation :

* Phase 1

  * ESS
  * BMI
  * Questionnaire : Nottingham health profile
  * Comorbidities -medical therapy
  * Smoking/alcohol Consumption
  * Then, we give an Actigraph (Body Media Sense WearÒ) to the patients, that he has to wear during 7 complete days
* Phase 2

  * Actigraphy report
  * Start of CPAP therapy(pressure adjusted according to autoCPAP device report after minimum one night)

Second Evaluation, after 3 months under CPAP:

* Phase 1

  § ESS
* BMI
* CPAP observance report to calculate mean use/day
* Questionnaire : Nottingham health profile
* Actigraph (Body Media Sense WearÒ) to the patients, that he has to wear during 7 complete days
* Phase 2: after 1 week under CPAP and actigraphy

  * Actigraphy report
  * CPAP observance report
  * CPAP Tolerance Questionnaire Ø

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe OSA
* sleepy (sleepiness assessed by Epworth Sleepiness Scale)
* indication for CPAP therapy

Exclusion Criteria:

* narcolepsy
* age < 18
* non sleepy Moderate to severe OSA
* no CPAP treatment required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe OSA
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU St Pierre, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obstructive Sleep Apnea, CPAP
Started | 150
Completed | 142
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Obstructive Sleep Apnea, CPAP
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 90
Region of Enrollment [Number; unit: participants]
  Belgium | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Sleep Time Before and After CPAP Therapy in Obstructive Sleep Apnea Patients
Description: change in Total sleep time before and after CPAP therapy in obstructive sleep apnea patients, assessed by actigraphy
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Obstructive Sleep Apnea, CPAP
Number analyzed (Participants) | 142
minutes | 29 (17)
Statistical Analysis 1: Comparison: Obstructive Sleep Apnea, CPAP; A power analysis conducted prior to the study predicted that a sample of 144 patients would provide an 80% power to detect a mean difference in sleep time of 40 minutes, assuming a standard deviation of 85 minutes and using a two-sided significance level of 5%; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Physical Activity (Number of Steps/Day)Before and After CPAP Therapy in OSA Patients
Description: Change in Physical activity (number of steps/day)before and after CPAP therapy in OSA patientsevaluated by actigraphy
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Obstructive Sleep Apnea, CPAP
Number analyzed (Participants) | 142
steps | 369 (157)
Statistical Analysis 1: Comparison: Obstructive Sleep Apnea, CPAP; Multiple regression modelling was used to determine whether actigraphic or polysomnographic data were predictors for physical activity, independently from age and BMI, stepwise forward selection of variables was performed; Test type: Superiority or Other; p < 0.05, Regression, Linear — Multiple regression modelling was used to determine whether actigraphic or polysomnographic data were predictors for physical activity, independently from age and BMI, stepwise forward selection of variables was performed

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Obstructive Sleep Apnea, CPAP
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes